CLINICAL TRIAL: NCT06683950
Title: Efficacy of Switching to Aflibercept 8mg in Patients with Neovascular AMD Showing Limited Response to Faricimab or Aflibercept 2mg
Brief Title: Switching to Aflibercept 8mg in Patients Showing Limited Response to Previous Treatment
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Kim's Eye Hospital (Other)
Responsible Party: Principal Investigator, Jae Hui Kim, Director of Clinical Research Center, Kim's Eye Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-07-002
Record Dates: First submitted 2024-10-27; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-10

CONDITIONS: Age-related Macular Degeneration (ARMD)
Keywords: Age-related macular degeneration; Choroidal neovascularization; Aflibercept; Aflibercept 8mg; Faricimab; Refractory
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Aflibercept 8mg (Experimental): In cases where patients previously treated with faricimab or aflibercept 2mg were switched to aflibercept 8mg
  Interventions: Drug: Aflibercept 8mg

INTERVENTIONS:
Drug: Aflibercept 8mg — Switching to intravitreal aflibercept 8mg in patients previously treated with faricimab or aflibercept 2mg.
  The dosing schedule is as follows.
  1. A single dose of 8mg aflibercept was administered to all patients
  2. After treatment 1, follow-up observations were conducted at the same intervals as previous treatments. If complete fluid resolution (no evidence of SRF or IRF) is observed, an additional dose of 8mg aflibercept is administered, extending the dosing intervals by two weeks each time.
  3. Up to three doses of 8mg aflibercept can be administered.
  4. If, after the administration of 8mg aflibercept, follow-up observations reveal remaining SRF or IRF, the study concludes without additional dosing.

SUMMARY:
The treatment landscape for neovascular AMD has evolved with various anti-VEGF agents since 2006. Ranibizumab initially led the way, but its limited efficacy in reducing retinal edema paved the way for aflibercept in 2011, which became globally popular for its effectiveness and safety. Yet, aflibercept did not fully meet all patients' needs. In 2019, brolucizumab showed promising anatomical results but had higher risks of inflammation, limiting its use. Faricimab, introduced in 2022, aimed for longer-lasting effects by targeting VEGF-A and angiopoietin 2. Though it required fewer injections, questions remain about its long-term efficacy compared to aflibercept.

Despite recent advancements, no agent has established itself as the new standard since aflibercept's introduction, leaving significant unmet needs. Aflibercept 8mg, approved in 2023, has shown promise by matching long-term visual outcomes of aflibercept 2mg with fewer injections and comparable safety. This study examines the effects of switching to aflibercept 8mg for patients with a limited response to previous treatments, addressing the potential for aflibercept 8mg to meet current needs more effectively and providing timely data for its global rollout.

DETAILED DESCRIPTION:
The treatment of neovascular AMD with anti-VEGF agents has evolved significantly. Introduced in 2006, ranibizumab heralded the era of anti-VEGF therapies but had limitations in duration and effectiveness in reducing retinal edema. To overcome these issues, aflibercept was introduced in 2011 and has been recognized for its superior efficacy and safety,1 becoming the most widely used drug globally. However, aflibercept also showed limited response in some patients, and the duration of its effectiveness was not always satisfactory.

Brolucizumab, introduced in 2019, demonstrated excellent anatomical outcomes but had a relatively high incidence of intraocular inflammation, ranging from 3 to 10%, preventing it from becoming a widely accepted standard treatment. The most recent, faricimab, introduced in 2022, was developed to inhibit not only VEGF-A but also angiopoietin 2, aiming for longer-lasting effects. In the TENAYA/LUCERNE clinical trials comparing its efficacy and safety with aflibercept, faricimab showed similar effects with fewer injections. However, due to differences in the treatment protocols between the aflibercept and faricimab groups, there remains a question about whether faricimab truly offers a longer duration of effect.

In conclusion, despite the introduction of brolucizumab and faricimab over the long span of 13 years since aflibercept was first introduced, these drugs have struggled to establish themselves as the new standard agents, especially when considering their overall efficacy and safety. Consequently, there has been a significant accumulation of unmet needs in the clinical treatment landscape over this extended period.

Aflibercept 8mg, the most recently FDA-approved agent in 2023, demonstrated not only superior initial anatomical effects compared to aflibercept 2mg in the PULSAR study, but also achieved similar long-term visual outcomes with fewer injections. Furthermore, it exhibited excellent safety, comparable to that of aflibercept 2mg. Based on these outcomes, many experts anticipate that aflibercept 8mg will become the new standard agent in the treatment of neovascular AMD, officially succeeding aflibercept 2mg.

Excluding aflibercept 2mg, faricimab could be considered the strongest contender for establishing aflibercept 8mg as the new standard. This is attributed to faricimab demonstrating satisfactory effects and excellent safety in clinical trials, as well as in subsequent real-world studies. Currently, there are no head-to-head clinical trials comparing these two drugs, and even if such trials are planned, it would take a considerable amount of time to ascertain the results. However, there is a simpler method to compare the effectiveness of a new agent against existing ones, which involves evaluating the effects of switching treatment in patients who have shown limited response to the current medication. In fact, such switching to new pharmaceutical agents after their introduction is widely practiced in clinical settings.10 Historically, the excellent efficacy observed when switching from ranibizumab to aflibercept 2mg played a significant role in the widespread adoption of aflibercept 2mg.

In this study, investigators aimed to evaluate the effects of switching to aflibercept 8mg in patients who have shown limited response to previous faricimab or aflibercept 2mg treatment. To the best of our knowledge, no such study has been reported in the English literature so far. This study not only has the potential to highlight the extended duration of action of aflibercept 8mg, but also holds significant importance in addressing the current unmet needs in the treatment of neovascular AMD. Additionally, by completing the study in a short period, investigators can contribute to generating timely data that aligns with the global introduction of aflibercept 8mg.

ELIGIBILITY:
Inclusion Criteria:

* Willing, committed, and able to return for ALL clinic visits and complete all study related procedures.
* Able to read, (or, if unable to read due to visual impairment, be read to verbatim by the person administering the informed consent or a family member) understand and willing to sign the informed consent form.
* Signed informed consent
* Patients aged 50 years or older
* Patients diagnosed with neovascular AMD or PCV
* Patients underwent faricimab or aflibercept 2mg injections with an inverval of 4 to 16 weeks
* Patients who continued to show persistent subretinal fluid (SRF) or intraretinal fluid (IRF) despite receiving two consecutive faricimab or aflibercept 2mg injections at the same injection interval.
* In cases where the central retinal thickness did not decrease by more than 50 μm during two consecutive treatments prior to inclusion in the study
* ETDRS BCVA letter score ≥25 letters (approximately 20/320 or better) in the study eye

Exclusion Criteria:

* Any prior ocular (in the study eye) or systemic treatment or surgery for neovascular AMD except dietary supplements or vitamins.
* Significant media opacities, including cataract, in the study eye that might interfere with visual acuity, assessment of safety, or fundus photography.
* Any concurrent ocular condition in the study eye which, in the opinion of the investigator, could either increase the risk to the patient beyond what is to be expected from standard procedures of intraocular injection, or which otherwise may interfere with the injection procedure or with evaluation of efficacy or safety.
* Any ocular or periocular infection within the last 2 weeks prior to Screening in either eye.
* Any history of uveitis in either eye.
* Presence of definite chorioretional anastomosis
* Scar or fibrosis, making up > 50% of total lesion in the study eye.
* Scar, fibrosis, or atrophy involving the center of the fovea in the study eye.
* Presence of retinal pigment epithelial tears or rips involving the macula in the study eye.
* History or clinical evidence of diabetic retinopathy, diabetic macular edema or any other vascular disease affecting the retina, other than AMD, in either eye.
* Any concurrent intraocular condition in the study eye (e.g. cataract) that, in the opinion of the investigator, could require either medical or surgical intervention during the 76 week study period.
* Prior vitrectomy in the study eye
* Any history of macular hole of stage 2 and above in the study eye.
* Any intraocular or periocular surgery within 3 months of Day 1 on the study eye, except lid surgery, which may not have taken place within 1 month of day 1, as long as its unlikely to interfere with the injection.
* Prior trabeculectomy or other filtration surgery in the study eye.
* Uncontrolled glaucoma (defined as intraocular pressure ≥ 25 mmHg despite treatment with antiglaucoma medication) in the study eye.
* Active intraocular inflammation in either eye.
* Active ocular or periocular infection in either eye.
* Aphakia or pseudophakia with absence of posterior capsule (unless it occurred as a result of a yttrium aluminum garnet [YAG] posterior capsulotomy) in the study eye.
* History of corneal transplant or corneal dystrophy in the study eye.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Presence of retinal fluid | Between 8 - 16 weeks (At the same interval as the previous dosing schedule for aflibercept 2mg or faricimab)
  To access changes in retinal fluid after switching to aflibercept 8mg in patients who showed limited response to faricimab or aflibercept 2mg treatment in neovascular AMD

SECONDARY OUTCOMES:
Change in best-corrected visual acuity (BCVA) | Between 8 - 16 weeks (At the same interval as the previous dosing schedule for aflibercept 2mg or faricimab)
  Change in best-corrected visual acuity (BCVA) after the switching to aflibercept 8mg
Change in central retinal thickness (CRT) | Between 8 - 16 weeks (At the same interval as the previous dosing schedule for aflibercept 2mg or faricimab)
  Change in central retinal thickness (CRT) after switching to aflibercept 8mg
Change in subfoveal choroidal thickness (SCT) | Between 8 - 16 weeks (At the same interval as the previous dosing schedule for aflibercept 2mg or faricimab)
  Change in subfoveal choroidal thickness (SCT) after switching to aflibercept 8mg
Change in the size of neovascularization | Between 8 - 16 weeks (At the same interval as the previous dosing schedule for aflibercept 2mg or faricimab)
  Change in the size of neovascularization as measured by OCT-A following the switching
Maximum fluid-free period | Between 8 - 16 weeks (At the same interval as the previous dosing schedule for aflibercept 2mg or faricimab or 2 weeks longer or 4 weeks longer)
  The longest fluid-free period (in weeks) maintained after switching to aflibercept 8mg, as assessed by optical coherence tomography images.
The proportion of eyes exhibiting fluid | Between 8 - 16 weeks (At the same interval as the previous dosing schedule for aflibercept 2mg or faricimab)
  The proportion of eyes exhibiting SRF, IRF, and PED

CONTACTS AND LOCATIONS:
Locations (1):
- Kim's Eye Hospital, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lanzetta P, Korobelnik JF, Heier JS, Leal S, Holz FG, Clark WL, Eichenbaum D, Iida T, Xiaodong S, Berliner AJ, Schulze A, Schmelter T, Schmidt-Ott U, Zhang X, Vitti R, Chu KW, Reed K, Rao R, Bhore R, Cheng Y, Sun W, Hirshberg B, Yancopoulos GD, Wong TY; PULSAR Investigators. Intravitreal aflibercept 8 mg in neovascular age-related macular degeneration (PULSAR): 48-week results from a randomised, double-masked, non-inferiority, phase 3 trial. Lancet. 2024 Mar 23;403(10432):1141-1152. doi: 10.1016/S0140-6736(24)00063-1. Epub 2024 Mar 7. PMID 38461841
- [Background] Wykoff CC, Brown DM, Reed K, Berliner AJ, Gerstenblith AT, Breazna A, Abraham P, Fein JG, Chu KW, Clark WL, Leal S, Schmelter T, Hirshberg B, Yancopoulos GD, Vitti R; CANDELA Study Investigators. Effect of High-Dose Intravitreal Aflibercept, 8 mg, in Patients With Neovascular Age-Related Macular Degeneration: The Phase 2 CANDELA Randomized Clinical Trial. JAMA Ophthalmol. 2023 Sep 1;141(9):834-842. doi: 10.1001/jamaophthalmol.2023.2421. PMID 37535382
- [Background] Raimondi R, Felfeli T, Bogdanova-Bennet A, Varma D, Habib M, Kotagiri A, Steel DH, Grinton M. Outcomes of Treatment-Resistant Neovascular Age-Related Macular Degeneration Switched from Aflibercept to Faricimab. Ophthalmol Retina. 2024 Jun;8(6):537-544. doi: 10.1016/j.oret.2023.11.015. Epub 2023 Nov 29. PMID 38040055
- [Background] Wijesingha N, Sivaprasad S. Infographic: Efficacy, durability, and safety of intravitreal faricimab up to every 16 weeks for neovascular age-related macular degeneration (TENAYA and LUCERNE). Eye (Lond). 2024 Aug;38(Suppl 2):53-54. doi: 10.1038/s41433-023-02867-4. Epub 2023 Dec 20. No abstract available. PMID 38123670
- [Background] Heier JS, Brown DM, Chong V, Korobelnik JF, Kaiser PK, Nguyen QD, Kirchhof B, Ho A, Ogura Y, Yancopoulos GD, Stahl N, Vitti R, Berliner AJ, Soo Y, Anderesi M, Groetzbach G, Sommerauer B, Sandbrink R, Simader C, Schmidt-Erfurth U; VIEW 1 and VIEW 2 Study Groups. Intravitreal aflibercept (VEGF trap-eye) in wet age-related macular degeneration. Ophthalmology. 2012 Dec;119(12):2537-48. doi: 10.1016/j.ophtha.2012.09.006. Epub 2012 Oct 17. PMID 23084240